CLINICAL TRIAL: NCT05270746
Title: The Predictive Value of Retinal Vascular Signs for Patients With Intracranial Artery Stenosis: A Prospective, Continuity Study, Cross-sectional Study
Brief Title: The Predictive Value of Retinal Vascular Signs for Intracranial Artery Stenosis (RVS-ICAS)
Acronym: RVS-ICAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Other Study IDs: RVS-ICAS
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Intracranial Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intracranial artery stenosis (ICAS) is a leading cause of ischemic stroke worldwide, contributing to the global burden of stroke, particularly in the Asian population. However, there is no non-invasive, easy to popularize and economic for intracranial artery stenosis in mass population screening. This study aims to evaluate the predictive value of retinal vascular signs for intracranial artery stenosis (ICAS) and explore a new screening method.

DETAILED DESCRIPTION:
Intracranial atherosclerosis stenosis (ICAS) is a leading cause of ischemic stroke worldwide, contributing to the global burden of stroke, particularly in the Asian population. Compared with the other stroke subtypes, patients with ICAS particularly the degree of stenosis≥50% had more severe stroke, stayed longer in the hospital and higher risk of recurrent ischemic events. However, there is no non-invasive, easy to popularize and economic for intracranial artery stenosis in mass population screening. Retinal imaging has great advantages including share the same embryological origin, anatomic features, and physiological properties with brain, non-invasive, easy to popularize, inexpensive and possess good economic benefits. Therefore, investigators design this study to assess the predictive value of retinal vascular signs for intracranial artery stenosis (ICAS) and hope to explore a new screening method.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥35
2. Accept TCD examination and fundus examination
3. Signed informed consent

Exclusion Criteria:

1. Non-atherosclerotic stenosis, such as arteritis, moyamoya disease, arterial dissection, vascular malformation, etc., which were clearly diagnosed.
2. Intracranial space-occupying lesions
3. Jugular vein and intracranial venous lesions
4. Patients with severe cardiac, hepatic, renal disease.
5. Life expectancy of less than 1 year due to co-morbid conditions.
6. Known pregnancy (or positive pregnancy test), or breast-feeding.
7. Pathological myopia fundus changes
8. Glaucoma
9. Refractive medium turbidity affects fundus observation
10. Anterior macular membrane of both eyes
11. Papilledema, optic neuritis and optic neuropathy
12. Patients who have had internal eye surgery in the last six months (including fundus laser)
13. Previous history of internal eye trauma
14. Poor image quality of fundus and images
15. Any condition which, in the judgment of the investigator, might increase the risk to the patient.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmic consultation center
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-27 (Estimated); Primary Completion 2022-06-26 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 6 months
  Number of true positives /(number of true positives + number of false negatives)*100
Specificity | 6 months
  Number of true negatives /(number of true negatives + number of false positives)*100
Positive predictive value | 6 months
  Positive predictive value = true positive cases /(true positive cases + false positive cases)*100
Negative predictive value | 6 months
  Negative predictive value = number of true negatives /(number of true negatives + number of false negatives)*100

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Fengtai District
  - Xuanwu hospital;Capital Medical University, Beijin, XI Cheng District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmstedt CA, Turan TN, Chimowitz MI. Atherosclerotic intracranial arterial stenosis: risk factors, diagnosis, and treatment. Lancet Neurol. 2013 Nov;12(11):1106-14. doi: 10.1016/S1474-4422(13)70195-9. PMID 24135208
- [Background] Wang Y, Zhao X, Liu L, Soo YO, Pu Y, Pan Y, Wang Y, Zou X, Leung TW, Cai Y, Bai Q, Wu Y, Wang C, Pan X, Luo B, Wong KS; CICAS Study Group. Prevalence and outcomes of symptomatic intracranial large artery stenoses and occlusions in China: the Chinese Intracranial Atherosclerosis (CICAS) Study. Stroke. 2014 Mar;45(3):663-9. doi: 10.1161/STROKEAHA.113.003508. Epub 2014 Jan 30. PMID 24481975
- [Background] Waters MF, Hoh BL, Lynn MJ, Kwon HM, Turan TN, Derdeyn CP, Fiorella D, Khanna A, Sheehan TO, Lane BF, Janis S, Montgomery J, Chimowitz MI; Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis (SAMMPRIS) Trial Investigators. Factors Associated With Recurrent Ischemic Stroke in the Medical Group of the SAMMPRIS Trial. JAMA Neurol. 2016 Mar;73(3):308-15. doi: 10.1001/jamaneurol.2015.4315. PMID 26747792
- [Background] Famakin BM, Chimowitz MI, Lynn MJ, Stern BJ, George MG; WASID Trial Investigators. Causes and severity of ischemic stroke in patients with symptomatic intracranial arterial stenosis. Stroke. 2009 Jun;40(6):1999-2003. doi: 10.1161/STROKEAHA.108.546150. Epub 2009 Apr 30. PMID 19407228
- [Background] London A, Benhar I, Schwartz M. The retina as a window to the brain-from eye research to CNS disorders. Nat Rev Neurol. 2013 Jan;9(1):44-53. doi: 10.1038/nrneurol.2012.227. Epub 2012 Nov 20. PMID 23165340
- [Background] Cheung CY, Ikram MK, Chen C, Wong TY. Imaging retina to study dementia and stroke. Prog Retin Eye Res. 2017 Mar;57:89-107. doi: 10.1016/j.preteyeres.2017.01.001. Epub 2017 Jan 3. PMID 28057562